CLINICAL TRIAL: NCT02204943
Title: Pharmacodynamic Study of Radium-223 in Men With Bone Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00053925
Record Dates: First submitted 2014-07-28; First posted 2014-07-31 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Bone Metastatic Castration-Resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Bone Biopsy and Circulating Tumor Cell Samples (Experimental)
  Interventions: Device: Biomarker analysis; Drug: Administration of radium-223

INTERVENTIONS:
Device: Biomarker analysis — Pharmacodynamic study of Radium-223 in bone biopsy and circulating tumor cell samples
Drug: Administration of radium-223 — Subjects will receive radium-223 treatment for their disease as standard of care in this protocol. They will be receiving this treatment regardless of their participation in this protocol.

SUMMARY:
This study will examine biomarkers involved in osteomimicry in bone metastases and circulating tumor cells (CTCs) of men with mCRPC before and during therapy with the bone-targeting radiopharmaceutical radium-223. This study will also examine the bio-distribution of radium-223 in bone and bone metastases of men with mCRPC.

The investigators hypothesize that bone metastases and CTCs in men with mCRPC will commonly express markers of EMT/plasticity and osteomimicry, not just in the normal surrounding osteoblastic stroma but in the epithelial tumor cells themselves and that radium-223 will target both of these compartments including the more mesenchymal/osteoblastic tumor cells and the surrounding osteoblasts in the active bone microenvironment, with a relative sparing of normal bone and bone marrow.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Life expectancy of at least 12 weeks (3 months).
3. Subjects must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.
4. Histologically confirmed diagnosis of adenocarcinoma of the prostate. Histologic variants of prostate cancer, including neuroendocrine features are permitted; however, pure small cell carcinoma of the prostate is excluded.
5. Presence of >2 sites of metastatic disease in bone as determined by bone scan or CT, and for men who opt-in for bone biopsy, they must have at least one site amenable to radiographically-guided metastatic biopsy as determined by the study radiologist.
6. Symptomatic castration-resistant bone metastatic disease as determined by the provider.
7. Prior or concurrent therapy with either abiraterone acetate or enzalutamide.
8. Ongoing ADT using an LHRH agonist (e.g. leuprolide, goserelin) or antagonist (e.g. degarelix) must continue on therapy unless prior bilateral orchiectomy has been performed.
9. Current evidence of disease progression as evidenced by one of the following:

   1. 2 consecutive rising PSA levels separated at least 1 week apart above nadir PSA on last systemic therapy. If no nadir, then 2 rising PSA values greater than baseline pretreatment value is required from the most immediate prior therapy, OR
   2. CT or bone scan based evidence of disease progression with bone metastasis (new lesions or growth of existing lesions), OR
   3. Evidence of symptomatic progression (increased pain in an area with known lesions confirmed on imaging).
10. All acute toxic effects of any prior treatment have resolved to NCI-CTCAE v4.0 Grade 2 or less.
11. Men of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 30 days after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate.
12. Acceptable hematology and serum biochemistry screening values:

    * White Blood Cell Count (WBC) ≥ 3,000/mm3
    * Absolute Neutrophil Count (ANC) ≥ 1,500/mm3
    * Platelet (PLT) count ≥ 100,000/mm3
    * Hemoglobin (HGB) ≥ 9.0 g/dl
    * Total bilirubin level ≤ 1.5 x institutional upper limit of normal (ULN)
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
    * Creatinine ≤ 1.5 x ULN
    * Albumin > 2.5 g/dL
13. Willing and able to comply with the protocol, including follow-up visits and examinations

Exclusion Criteria:

1. Treatment with cytotoxic chemotherapy within previous 4 weeks, or failure to recover from AEs down to grade 2 or less due to cytotoxic chemotherapy administered more than 4 weeks previous (however, ongoing neuropathy is permitted)
2. Receiving concurrent systemic therapy with radionuclides (e.g., strontium-89, samarium-153, rhenium-186, or rhenium-188) for the treatment of bony metastases. Prior therapy with radium-223 is not permitted.
3. Other malignancy treated within the last 3 years (except non melanoma skin cancer or low-grade superficial bladder cancer)
4. Visceral (i.e. liver, lung, etc) metastases (pulmonary nodules ≤1cm are permitted) as assessed by chest, abdominal or pelvic computed tomography (CT) (or other imaging modality)
5. Presence of active untreated CNS parenchymal or epidural spinal metastases
6. Lymphadenopathy exceeding 3 cm in short-axis diameter
7. Imminent spinal cord compression based on clinical findings and/or magnetic resonance imaging (MRI). Treatment should be completed for spinal cord compression.
8. Any other serious illness or medical condition, such as but not limited to:

   * Any infection ≥ National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0 Grade 2
   * Cardiac failure New York Heart Association (NYHA) III or IV
   * Crohn's disease or ulcerative colitis
   * Bone marrow dysplasia
   * Fecal incontinence
9. Inability to comply with the protocol and/or not willing or not available for follow-up assessments.
10. Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
11. Concurrent cytotoxic chemotherapy or anticancer therapies other than abiraterone, prednisone or other glucocorticoids, enzalutamide, androgen deprivation therapy, bisphosphonates, and denosumab.
12. Concurrent use of another investigational drug or device therapy (i.e., outside of study treatment) during, or within 2 weeks of treatment initiation.
13. Major surgery within 30 days prior to start of study drug.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who overexpress alkaline phosphatase (ALP) in Circulating Tumor Cells (CTCs) at each time point | Cycle 1 Day 1, Cycle 3 Day 1 and Cycle 6 Day 1 or disease progression
  The proportion of patients who over-express ALP in the CTCs, defined as any over-expression, will be estimated using descriptive statistics at each time point. ALP expression will be concurrently examined in the bone metastatic biopsies of men as well, if evaluable tissue is available.

SECONDARY OUTCOMES:
Change in biomarkers of epithelial plasticity and osteomimicry expressed in the bone metastases of men with bone metastatic CRPC | At time of optional biopsy, pre- and post-treatment with Radium-223. Post-treatment biopsies will be approximately 10 and 22 weeks after first treatment.
  Summary statistics of other biomarkers involved in epithelial plasticity and osteomimicry in the tumor tissue of men with bone metastatic CRPC including expression of ALP, PSA, CK, O-cadherin, N-cadherin, vimentin, TWIST, SNAIL, beta-catenin, ZEB1, androgen receptor (AR), AR variants (ARv) and γ-H2AX will be completed.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Armstrong, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Armstrong AJ, Gupta S, Healy P, Kemeny G, Leith B, Zalutsky MR, Spritzer C, Davies C, Rothwell C, Ware K, Somarelli JA, Wood K, Ribar T, Giannakakou P, Zhang J, Gerber D, Anand M, Foo WC, Halabi S, Gregory SG, George DJ. Pharmacodynamic study of radium-223 in men with bone metastatic castration resistant prostate cancer. PLoS One. 2019 May 28;14(5):e0216934. doi: 10.1371/journal.pone.0216934. eCollection 2019. PMID 31136607